CLINICAL TRIAL: NCT04875793
Title: Effectiveness of an Integrated Colorectal Cancer Screening System in Saudi Arabia: A Pragmatic Randomized Trial
Brief Title: Effectiveness of an Integrated Colorectal Cancer Screening in Saudi Arabia: A Pragmatic Randomized Trial
Acronym: CRCScreen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tabuk (Other)
Collaborators: Ein Al-Hayat Medical Complex (Unknown); The Charitable Society for Health Care in Tabuk (Unknown); Ministry of Health, Saudi Arabia (Other Government); Vision Health Consultancy Firm, Sudan (Unknown)
Responsible Party: Principal Investigator, Fakhralddin Abbas Mohammed Elfakki, Assistant Professor of Preventive Medicine and Epidemiology, University of Tabuk
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TU-077/019/012
Record Dates: First submitted 2021-05-01; First posted 2021-05-06 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Neoplasms; Colorectal Cancer; Colonic Polyp; Occult Bleeding
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps | interventions — Defecation; Occult Blood; Colonoscopy

STUDY DESIGN:
Intervention Model Description: List of health centres that randomly allocated to receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- List of health centers that randomly allocated to receive the intervention (Experimental): The intervention is the integrated system which is composed of psychologist, endoscopy physician, family physician, community outreach, and audiovisuals in the waiting area. In addition to text messages of information, education and communication (IEC) delivered to the participants at the outreach, and education campaigns to mobilize individuals going for screening.
  Interventions: Diagnostic Test: Stool for Occult Blood Test and Colonoscopy with comprehensive medical checkups
- List of health centers that randomly allocated to receive routine care (No Intervention): The comparators will be individuals with an average risk of colorectal cancer of both genders attending the randomly selected health centres

INTERVENTIONS:
Diagnostic Test: Stool for Occult Blood Test and Colonoscopy with comprehensive medical checkups — participants will be drawn from all public government institutions inside Tabuk city(outreach). The institution head will be requested to give wellness cards to the eligible employee to receive comprehensive testing for free in addition to CRC test in selected public health centres.
  Other Names: Facilitated appointment to receive a digestive health check and a comprehensive medical checkups
  Arms: List of health centers that randomly allocated to receive the intervention

SUMMARY:
The global burden of colorectal cancer (CRC) incidence among young age groups is rising and overwhelming. This new trend of young-onset CRC incidence is evident in western countries. Unfortunately, Asian countries have shown the same epidemic shift in the past few years. As a consequence, this situation might necessitate revisiting the current screening program in this region.

Saudi Arabia has a two-fold increase in CRC incidence among young age groups in the last 18 years (9.6/100000 for male versus 9.3/100000 for female). This rising incidence ascribed to the lack of a screening program and suggested lowering CRC screening to 40.

The low awareness about risk factors, signs, and symptoms of the disease causes late presentation of CRC cases. Therefore, most presenting cases are associated with a poor prognosis and short survival. Educational and screening programs are, by no means, considered valuable and essential as CRC tends to affect younger age groups.

DETAILED DESCRIPTION:
CRC is cancer that starts in the innermost lining mucosa of the colon or rectum. According to the global cancer Observatory (GCO) 2018, CRC incidence is the third (10.2%) globally, after lung and breast cancers (11.6%). In Saudi Arabia, 2010 report, the incidence was 10.4/100,000 that slightly higher in male groups. Unfortunately, the incidence among young age groups is more than that in countries with high incidence.

Most of the CRCs initially found as small benign growth or projections known as polyps inside the lumen of colorectal space. A polyp is precancerous if it is >1 cm or the presence of more than two polyps, or if dysplasia present after the polyp removal. There are two main types of polyps: precancerous and hyperplastic polyps or inflammatory polyps, which are not precancerous. The early resection will prevent future cancer development and total cure.

Different lifestyle factors that could increase CRC's risk include lack of regular physical exercise, a diet low in fruit and vegetables, a low-fibre and high-fat diet, diary intake during adolescence, overweight and obesity, alcohol consumption and tobacco use. Adherence to CRC screening is essential to limit CRC cancer incidence and improve population health; and then, health providers need to understand the stages of the disease to recommend effective screening strategies.

ELIGIBILITY:
Inclusion Criteria:

* The participants will be individuals with an average risk of colorectal cancer, age: 40 years and above of both genders

Exclusion Criteria:

* Individuals age less than 40 years or severely ill individuals

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
The percentage of individuals who screened positive in the intervention group vs. control group. | 1 - 12 months
  The comparison of rate positive screening between the intervention and routine care
The enrollment rate of individuals who underwent CRC screening in the intervention group vs. control group | 1 - 12 months
  The comparison of the enrollment rate between the intervention and routine care

SECONDARY OUTCOMES:
The percentage of individuals who screened positive and enrolled in colonoscopy for follow-up in the intervention group vs. control group. | 1 - 12 months
  Per cent of enrollment in colonoscopy appointment and future follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Public Primary Health Care Centers in the Tabuk City, Tabuk, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol